CLINICAL TRIAL: NCT00179101
Title: Effect of Deep Brain Stimulation on Depression and Quality of Life in Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Other Study IDs: 040251
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Depression; Quality of Life; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Deep Brain Stimulation

SUMMARY:
We will evaluate the effect of deep brain stimulation on the depression and quality of life in Parkinson's disease. We aim to compare depression pre-operatively and post-operatively in Parkinson's patients with deep brain stimulation to Parkinson's patients evaluated and approved for deep brain stimulation but who did not complete surgery. We will also compare quality of life measures between patients with and without deep brain stimulation.

DETAILED DESCRIPTION:
Deep brain stimulation is an approved therapy for Parkinson's patients, and this procedure is actively performed at Vanderbilt University Hospital. Questions have been raised concerning the effect of deep brain stimulation on the depression commonly seen in Parkinson's patients. Through this study, we plan to evaluate and compare the incidence and severity of depression in Parkinson's patients with deep brain stimulation to those who did not complete the surgery. Primary literature has indicated a general increase in quality of life of those patients receiving DBS, but no studies have compared these two specific patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson's disease.
* Patients who have received neuropsychological testing in preparation for possible deep brain stimulation.
* Patients are within the age of 50 and 85.

Exclusion Criteria:

* Parkinson's patients not approved for deep brain stimulation on the basis of neuropsychological testing.
* Patients who received deep brain stimulation less than a year ago.
* Patients who do not consent to the study procedures.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-04; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Courtney R Schadt, BS, Principal Investigator — Vanderbilt University; David Charles, MD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States